CLINICAL TRIAL: NCT01203254
Title: Colesevelam for the Treatment of Bile Acid Malabsorption in Patients With Crohn's Disease
Acronym: COBAM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Florian Beigel (Other)
Responsible Party: Sponsor-Investigator, Florian Beigel, Dr. med., Klinikum der Universitaet Muenchen, Grosshadern
Organization: Klinikum der Universitaet Muenchen, Grosshadern (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-010727-91
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Crohns Disease; Bile Acid Malabsorption
Keywords: Colesevelam; IBD; Bile Acid Malabsorption; Crohns disease
MeSH Terms: conditions — Crohn Disease | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cholestagel (Active Comparator)
  Interventions: Drug: Colesevelam

INTERVENTIONS:
Drug: Colesevelam — Colesevelam 625 mg tablet; 3 times daily 2 tablets
  Arms: Cholestagel
Drug: Placebo — Placebo tablet: 3 times daily 2 tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of cholestagel to reduce the frequency of soft and liquid stools per day in patients with CD in clinical remission with symptoms of BAM and to assess the improvement in stool consistency and quality of life in these patients and to assess the safety of cholestagel.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent after adequate explanation of the patient information.
* Male and female patients with CD and 18 to 65 years of age in clinical remission with a Crohns Disease Activity Index (CDAI) score of 150 or less, with symptoms of functional BAM or symptoms of BAM after small bowel resection with a frequency of at least 3 to maximal 15 liquid or soft stools per day.
* Stable medical treatment of CD for a minimal period of 3 months preceding the screening visit, consisting of

  * either continuous oral treatment of aminosalicylate, prednisolone (a maximum 10 mg/day), azathioprine, 6-mercaptopurine, or methotrexate
  * or supporting periodic treatment* with TNF-alpha AK (Infliximab, Adalimumab, Certolizumab) (for patients on TNF-alpha, dosing with TNF-alpha should coincide with baseline visit)
* Blood serum CRP value of less or equal then 1 mg/dl (10 mg/l).
* BAM assessed with a blood test on a 7α-hydroxy-4-cholesten-3-on excretion of equal or more than 50 ng/ml

Exclusion criteria:

* Allergy or hypersensitivity to any of the components of cholestagel or placebo as identified from the medical history
* Participation at another clinical trial within a period of 4 weeks before the screening visit
* Presence of any addiction, alcohol abuse or specific disease that would not allow the patient to understand the essence and requirements and potential consequences of the participation to the clinical trial
* Signs suggestive of the patient being unable to follow the visit schedule as required (for example for professional obligations)
* Treatment with cyclosporine, or tacrolimus, 3 month or less before screening
* Oral Treatment with antibiotics 3 weeks or less before screening
* Topical treatment with steroid- or mesalazine-containing applications 3 weeks or less before screening
* Treatment with bile acid bile acid binding agent (e.g. Cholestayramine)6 weeks or less before screening
* Infectious diseases (HIV, hep B, hep C, tuberculosis, listeriosis, positive clostridium-difficile-toxin- proof in faeces)
* Current presence of intra-abdominal abscess or Fistula
* Cholestatic liver disease, bowel or biliary obstruction
* Dysphagia or swallowing disorders
* Known malignancy or history of malignancy
* Having undergone intestinal surgery within 6 months from screening
* Status after intestinal surgery with more then 100cm of resected bowel.
* Short bowel syndrome
* Planned -gastrostomy, ileostomy or colostomy.
* Pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Reduction of fluid stool > 30 % | 4 weeks after baseline

SECONDARY OUTCOMES:
Improvement of Stool Consistency | 4 weeks after baseline
  Proportion of patients on cholestagel compared to placebo that reaches improvement of stool consistency on the Bristol stool chart of at least one point.
Improvement of Quality of Life. | 4 weeks after baseline
  Proportion of patients on cholestagel compared to placebo that reaches an improvement of the Quality of Life.
Change of median liquid or soft stool frequency/per day. | 4 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Florian Beigel, M.D., Principal Investigator — Klinikum der Universität München - Grosshadern
Locations (6):
- Germany (6):
  - Praxis Dr. Mroß, Berlin
  - Hochschulambulanz Med. Klinik I - Charite-, Berlin
  - Hamburgisches Forschungsinstitut für CED, Hamburg
  - Universitätsklinikum des Saarlandes -Innere Medizin-, Homburg
  - Internistische Gemeinschaftspraxis, Leipzig
  - CED - Zentrum der Universität München - Klinikum Grosshadern, Munich

REFERENCES:
- [Derived] Beigel F, Teich N, Howaldt S, Lammert F, Maul J, Breiteneicher S, Rust C, Goke B, Brand S, Ochsenkuhn T. Colesevelam for the treatment of bile acid malabsorption-associated diarrhea in patients with Crohn's disease: a randomized, double-blind, placebo-controlled study. J Crohns Colitis. 2014 Nov;8(11):1471-9. doi: 10.1016/j.crohns.2014.05.009. Epub 2014 Jun 19. PMID 24953836